CLINICAL TRIAL: NCT00894777
Title: Management of Patients With Moderate and Severe Psoriasis Under Treatment With Topical and/or Systemic Drugs
Brief Title: Study Evaluating Management of Patients With Moderate and Severe Psoriasis
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Other Study IDs: 0881A6-4577
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with moderate and severe psoriasis under treatment with topical and/or systemic drugs
  Interventions: Other: Clinical record review

INTERVENTIONS:
Other: Clinical record review

SUMMARY:
This is an observational, naturalistic, multicenter, retrospective study to describe the therapeutic management of patients with moderate and severe psoriasis under treatment with topical and/or systemic drugs in usual clinical practice in Spain.

ELIGIBILITY:
Main Inclusion Criteria:

·Over 18 years of age.·Diagnosed with moderate or severe psoriasis.·Initiated treatment with topical and/or systemic treatment between two and five years before enrollment in the study. ·Has a clinical record at the dermatologist office.

Main Exclusion Criteria:

·Currently participating in a clinical study. ·Clinical record lacks minimum data required for observational analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate and severe psoriasis under treatment with topical and/or systemic drugs in usual clinical practice
Sampling Method: Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of the therapeutic management of patients with moderate and severe psoriasis under treatment with topical and/or systemic drugs including sequence, doses and duration of treatment. | 4 months

SECONDARY OUTCOMES:
Comparison of therapeutic management depending on patients' disease severity, using absolute and relative frequencies for qualitative variables and centralization and dispersion measures (mean, SD, median, minimum, maximum..) for quantitative variables. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Madrid, Madrid, Spain